CLINICAL TRIAL: NCT04211909
Title: A Phase 3b Multicenter, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/Velpatasvir Fixed-Dose Combination and Sofosbuvir/Velpatasvir/Voxilaprevir Fixed-Dose Combination for 12 Weeks in Subjects With Chronic HCV Infection
Brief Title: Study to Investigate the Efficacy and Safety of Sofosbuvir/Velpatasvir (SOF/VEL) Fixed-Dose Combination (FDC) and Sofosbuvir/Velpatasvir/Voxilaprevir (SOF/VEL/VOX ) FDC for 12 Weeks in Adults With Chronic Hepatitis C Virus (HCV) Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-342-5532
Record Dates: First submitted 2019-12-23; First posted 2019-12-26 (Actual); Results first posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-09

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination; sofosbuvir velpatasvir voxilaprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- SOF/VEL (Experimental): Participants with chronic HCV infection (genotype 1 or 2), who are treatment-naive or treatment-experienced with interferon (IFN)-based treatments will receive SOF/VEL for 12 weeks.
  Interventions: Drug: SOF/VEL
- SOF/VEL/VOX (Experimental): Participants with chronic HCV infection (genotype 1), who are treatment-experienced with nonstructural protein 5A (NS5A) direct-acting antiviral (DAA)-based treatments of at least 4 weeks duration will receive SOF/VEL/VOX for 12 weeks.
  Interventions: Drug: SOF/VEL/VOX

INTERVENTIONS:
Drug: SOF/VEL — 400/100 mg FDC tablet orally once daily.
  Other Names: Epclusa®; GS-7977/GS-5816
  Arms: SOF/VEL
Drug: SOF/VEL/VOX — 400/100/100 mg FDC tablet orally once daily.
  Other Names: Vosevi ®; GS-7977/GS-5816/GS-9857
  Arms: SOF/VEL/VOX

SUMMARY:
The primary objectives of this study are to evaluate the antiviral efficacy, safety, and tolerability of therapy with Sofosbuvir/Velpatasvir (SOF/VEL) Fixed-Dose Combination (FDC) and Sofosbuvir/Velpatasvir/Voxilaprevir (SOF/VEL/VOX ) FDC in participants with chronic HCV infection.

ELIGIBILITY:
Key Inclusion Criteria:

* Chronic HCV infected males and non-pregnant/non-lactating females
* Treatment-naive or treatment-experienced individuals
* Non-cirrhosis or compensated cirrhosis at screening

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (22):
- South Korea (22):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-D
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chosun University Hospital, Gwangju
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - VHS (Veterans Health Service) Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul Saint Mary's Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan University Hospital, Ulsan
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in South Korea. The first participant was screened on 03 January 2020. The last study visit occurred on 12 November 2020.
Pre-assignment Details: 96 participants were screened.
Groups:
- SOF/VEL: Participants with chronic hepatitis C virus (HCV) infection (genotype 1 or 2), who were treatment-naive or treatment-experienced with interferon (IFN)-based treatments received sofosbuvir/velpatasvir (SOF/VEL) (400/100 mg) fixed-dose combination (FDC) tablet orally once daily for 12 weeks.
- SOF/VEL/VOX: Participants with chronic HCV infection (genotype 1 or 2), who were treatment-experienced with nonstructural protein 5A (NS5A) direct-acting antiviral (DAA)-based treatments of at least a 4 weeks duration received sofosbuvir/velpatasvir/voxilaprevir (SOF/VEL/VOX) (400/100/100 mg) FDC tablet orally once daily for 12 weeks.
Period: Overall Study
Arm/Group | SOF/VEL | SOF/VEL/VOX
Started | 54 | 33
Completed | 54 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of the study drug.
Groups:
- SOF/VEL: Participants with chronic HCV infection (genotype 1 or 2), who were treatment-naive or treatment-experienced with IFN-based treatments received SOF/VEL 400/100 mg FDC tablet orally once daily for 12 weeks.
- SOF/VEL/VOX: Participants with chronic HCV infection (genotype 1 or 2), who were treatment-experienced with NS5A DAA-based treatments of at least a 4 weeks duration received SOF/VEL/VOX 400/100/100 mg FDC tablet orally once daily for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | SOF/VEL | SOF/VEL/VOX | Total
Number analyzed (Participants) | 54 | 33 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 17 | 51
  >=65 years | 20 | 16 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 18 | 47
  Male | 25 | 15 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 54 | 33 | 87
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity Not Permitted: local regulators did not allow collection of ethnicity information.
  Participants
    Ethnicity: Not Hispanic or Latino | 53 | 33 | 86
    Ethnicity: Not Permitted | 1 | 0 | 1
Interleukin-28B gene (IL28b) Status [Number; unit: participants] — The CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 41 | 23 | 64
    CT | 13 | 9 | 22
    TT | 0 | 0 | 0
    Missing | 0 | 1 | 1
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 24 | 3 | 27
  ≥ 800,000 IU/mL | 30 | 30 | 60
Genotype [Count of Participants; unit: Participants] — 1 participant with Genotype 2 in SOF/VEL/VOX arm was included because of eligibility criteria deviation.
  Participants
    Genotype 1 | 27 | 32 | 59
    Genotype 2 | 27 | 1 | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) < Lower Limit of Quantification (LLOQ) 12 Weeks After Discontinuation of Study Treatment
Description: SVR12 was defined as HCV RNA < LLOQ (i.e., 15 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set included all enrolled participants who took at least 1 dose of study drug and had detectable HCV RNA at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL | SOF/VEL/VOX
Number analyzed (Participants) | 53 | 33
percentage of participants | 98.1 [89.9 to 100.0] | 100 [89.4 to 100]

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued the Study Drug Due to an Adverse Event
Time Frame: First dose date up to 12 weeks plus 30 days
Population: Safety Analysis Set included all participants who took at least 1 dose of the study drug.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL | SOF/VEL/VOX
Number analyzed (Participants) | 54 | 33
percentage of participants | 1.9 | 0

3. Secondary Outcome: Percentage of Participants With SVR < LLOQ 4 Weeks After Discontinuation of Study Treatment
Description: SVR4 was defined as HCV RNA < LLOQ (i.e.15 IU/mL) 4 weeks after stopping study treatment.
Time Frame: Posttreatment Week 4
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SOF/VEL | SOF/VEL/VOX
Number analyzed (Participants) | 53 | 33
percentage of participants | 98.1 [89.9 to 100.0] | 100 [89.4 to 100]

4. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure was defined as:
  On-treatment virologic failure:
  * Breakthrough (HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ, while on treatment, confirmed with 2 consecutive values), or
  * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
  * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment )
  Virologic relapse:
  • Confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit
Time Frame: Baseline up to Posttreatment Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL | SOF/VEL/VOX
Number analyzed (Participants) | 53 | 33
percentage of participants | 1.9 | 0

5. Secondary Outcome: Percentage of Participants With HCV RNA < LLOQ on Treatment
Description: LLOQ was 15 IU/mL.
Time Frame: Week 2, Week 4, Week 8, Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | SOF/VEL | SOF/VEL/VOX
Number analyzed (Participants) | 53 | 33
percentage of participants
  Week 2 | 90.6 | 69.7
  Week 4 | 100.0 | 100.0
  Week 8: number analyzed (Participants) | 52 | 33
  Week 8 | 100.0 | 100.0
  Week 12: number analyzed (Participants) | 52 | 33
  Week 12 | 100.0 | 100.0

6. Secondary Outcome: Change From Baseline in HCV RNA
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | SOF/VEL | SOF/VEL/VOX
Number analyzed (Participants) | 53 | 33
log10 IU/mL
  Baseline | 5.95 (0.866) | 6.48 (0.354)
  Change at Week 2: number analyzed (Participants) | 52 | 33
  Change at Week 2 | -4.78 (0.857) | -5.19 (0.545)
  Change at Week 4: number analyzed (Participants) | 53 | 32
  Change at Week 4 | -4.81 (0.866) | -5.33 (0.354)
  Change at Week 8: number analyzed (Participants) | 52 | 33
  Change at Week 8 | -4.79 (0.867) | -5.33 (0.354)
  Change at Week 12: number analyzed (Participants) | 52 | 33
  Change at Week 12 | -4.79 (0.867) | -5.33 (0.354)

7. Secondary Outcome: Number of Participants With Alanine Aminotransferase (ALT) Normalization
Description: Number of participants with ALT normalization, defined as ALT > upper limit of normal (ULN) (ULN = 43 U/L) at baseline and ALT ≤ ULN, at each visit was presented.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: participants
Arm/Group | SOF/VEL | SOF/VEL/VOX
Number analyzed (Participants) | 53 | 33
participants
  Baseline (ALT>ULN) | 21 | 16
  Week 2 (ALT≤ ULN): number analyzed (Participants) | 21 | 16
  Week 2 (ALT≤ ULN) | 21 | 13
  Week 4 (ALT≤ ULN): number analyzed (Participants) | 21 | 16
  Week 4 (ALT≤ ULN) | 21 | 13
  Week 8 (ALT≤ ULN): number analyzed (Participants) | 21 | 16
  Week 8 (ALT≤ ULN) | 19 | 13
  Week 12 (ALT≤ ULN): number analyzed (Participants) | 21 | 16
  Week 12 (ALT≤ ULN) | 17 | 13

ADVERSE EVENTS:
Time Frame: From first dose date up to 12 weeks plus 30 days
Description: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- SOF/VEL/VOX: Participants with chronic HCV infection (genotype 1 or 2), who were treatment-experienced with NS5A-DAA based treatments of at least a 4 weeks duration received SOF/VEL/VOX 400/100/100 mg FDC tablet orally once daily for 12 weeks.
Arm/Group | SOF/VEL | SOF/VEL/VOX
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/33
Serious Adverse Events (participants affected / at risk) | 3/54 | 1/33
Other Adverse Events (participants affected / at risk) | 5/54 | 8/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=54) | SOF/VEL/VOX (N=33)
Haematochezia (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF/VEL (N=54) | SOF/VEL/VOX (N=33)
Nausea (Gastrointestinal disorders) | 2 | 3
Headache (Nervous system disorders) | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT04211909/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/09/NCT04211909/SAP_001.pdf